CLINICAL TRIAL: NCT04313751
Title: Reducing Cardiovascular Disease Risk in Perimenopausal Latinas: Pilot Study of a Multi-Component Intervention
Brief Title: Reducing Cardiovascular Disease Risk in Perimenopausal Latinas
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 19-2756; K23MD014767 (NIH)
Record Dates: First submitted 2020-03-16; First posted 2020-03-18 (Actual); Results first posted 2024-08-20 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-04

CONDITIONS: Cardiovascular Risk Factor; Health Behavior; Physical Activity; Self Efficacy; Vascular Stiffness
Keywords: Hispanic/Latina; Menopause; Cardiovascular disease
MeSH Terms: conditions — Health Behavior; Motor Activity; Cardiovascular Diseases | interventions — Educational Status; Exercise; Waiting Lists

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: After enrollment and baseline assessment, participants will be randomized to a community site receiving either the intervention or waitlist control.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Education, Physical Activity, and Stress Management Program (Experimental): Classes for the intervention group will be run by a bilingual interventionist and will last 120 minutes weekly for 12 weeks and then monthly for 3 months.
  Interventions: Behavioral: Education, Physical Activity, and Stress Management Program
- Wait-list Control (Active Comparator): Data in the wait-list control group will be collected at the same time intervals as the intervention group. After Time 3 data collection, they will be offered the Phase I intervention (12 weekly sessions).
  Interventions: Other: Wait-list

INTERVENTIONS:
Behavioral: Education, Physical Activity, and Stress Management Program — Twelve weekly classes for one hour focused on CVD risk factor education using the Su Corazón Su Vida curriculum and coping skills training followed by a 45 minute exercise class and 15 minute stress management session. Then they will return for one hour for continued support, a forty-five minute exercise class, and fifteen minute stress management session.
  Arms: Education, Physical Activity, and Stress Management Program
Other: Wait-list — The wait-list control group will receive 12 weekly one hour education and coping skills training sessions followed by a 45 minute exercise class and a 15 minute stress management session.
  Arms: Wait-list Control

SUMMARY:
The goal of this study is to pilot test a 12-week behavioral intervention among perimenopausal Latinas (age 40-55 years) that integrates evidence-based education with physical activity, stress management, and coping skills training to: 1) reduce cardiovascular disease (CVD) risk factors and arterial stiffness; 2) improve nutrition, physical activity, and sleep behaviors; and 3) improve stress management, coping strategies, and self-efficacy. This study will recruit participants from two community groups: one group will be randomly assigned to complete the intervention; the other will be a wait-list control.

DETAILED DESCRIPTION:
While CVD mortality is the leading cause of death in the United States, large racial/ethnic disparities in cardiovascular health exist between Latinas and non-Hispanic populations. Risk of CVD increases significantly for women following menopause. There are substantial increases in CVD risk factors during perimenopause, specifically, perimenopausal women exhibit greater visceral adipose tissue, fasting glucose, total cholesterol, and systolic blood pressure, compared to premenopausal women. Although behavioral intervention research targeting CVD risk during perimenopause emerged over the past decade, no studies were designed to decrease biological CVD risk among perimenopausal Latinas. This study will recruit perimenopausal Latinas (age 40-55 years) from two community groups: one group will be randomly assigned to complete the intervention; the other will be a wait-list control. This intervention has 3 phases: 12 weekly sessions (Phase I: education, physical activity, stress management, coping skills training) followed by 3 monthly sessions of continued support (Phase II); and finally 6 months of skill maintenance on their own (Phase III). Data will be collected at Time 1 (0 months [baseline]), Time 2 (6 months [completion of the intervention]) and Time 3 (12 months [after 6 months of maintenance on own]). Data collected will include biological CVD risk factors and arterial stiffness (primary outcomes: blood pressure, lipid profile, blood glucose, carotid-femoral pulse wave velocity). Secondary outcomes will include health behaviors and self-efficacy (Food Behavior Checklist, 7 day Accelerometer, Sleep Quality Scale, Eating Self-Efficacy Scale, Exercise Self-Efficacy Scale) and other biological factors related to CVD risk (waist circumference, weight, body mass index [BMI], C-reactive protein, hair cortisol). The investigators will also evaluate the feasibility of the intervention (e.g., enrollment and retention rates, barriers and facilitators to enrollment, intervention fidelity, suitability of study procedures and outcome measures, and participant satisfaction with the intervention and study protocol). The knowledge to be gained from this pilot study may provide a foundation for extending this intervention to a larger efficacy trial. This research holds potential to accelerate greatly the acquisition of knowledge related to CVD risk among perimenopausal Latinas, and the impact of behavioral interventions to reduce CVD risk in this underserved population.

ELIGIBILITY:
Inclusion Criteria:

* age 40-60 years
* self-identify as Hispanic/Latina
* understand spoken English or Spanish
* perimenopausal or early postmenopausal (menstrual bleeding in the past 3 months, but timing have varied in past year; no menstrual bleeding in the past 3-11 months; last menstrual cycle 12-24 months ago)
* intact uterus and at least one ovary
* not currently pregnant
* no hormone therapy or oral contraceptives in the past 3 months
* consent to join the study

Exclusion Criteria:

* heart murmur
* congenital heart disease
* family history of sudden death
* difficulty exercising
* history of CVD (heart attack, stroke, coronary heart disease)

Ages: 40 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 49 (Actual)
Dates: Start 2020-06-30 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yamnia I Cortes, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: At the close of the study and after the main data from the study has been published.
Access Criteria: Contact Dr. Yamnia I. Cortes at yicortes@email.unc.edu

REFERENCES:
- [Derived] Cortes YI, Harris LK, Cazales A, Marginean V, Long C, Woods-Giscombe CL, Perreira KM. Feasibility and acceptability of Menopausia, Salud, Corazon (Menopause, Health, Heart): a pilot randomized trial to reduce cardiovascular disease risk in midlife Latinas. Menopause. 2026 Feb 3. doi: 10.1097/GME.0000000000002718. Online ahead of print. PMID 41632258
- [Derived] Cortes YI, Duran M, Marginean V, Harris LK, Cazales A, Santiago L, Mislan MD, Perreira KM. Lessons Learned in Clinical Research Recruitment of Midlife Latinas During COVID-19. Menopause. 2022 Jul 1;29(7):883-888. doi: 10.1097/GME.0000000000001983. PMID 35796561
- [Derived] Cortes YI, Berry DC, Perreira KM, Stuebe A, Stoner L, Giscombe CW, Crandell J, Santiago L, Harris LK, Duran M. A multi-component, community-engaged intervention to reduce cardiovascular disease risk in perimenopausal Latinas: pilot study protocol. Pilot Feasibility Stud. 2021 Jan 6;7(1):10. doi: 10.1186/s40814-020-00756-1. PMID 33407947

RESULTS

PARTICIPANT FLOW:
Groups:
- Education, Physical Activity, and Stress Management Program: Classes for the intervention group will be run by a bilingual interventionist and will last 120 minutes weekly for 12 weeks and then monthly for 3 months.
  Education, Physical Activity, and Stress Management Program: Twelve weekly classes for one hour focused on cardiovascular disease (CVD) risk factor education using the Su Corazón Su Vida curriculum and coping skills training followed by a 45 minute exercise class and 15 minute stress management session. Then they will return for one hour for continued support, a forty-five minute exercise class, and fifteen minute stress management session.
Period: Overall Study
Arm/Group | Education, Physical Activity, and Stress Management Program | Wait-list Control
Started | 26 | 23
Completed | 21 | 16
Not Completed | 5 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Education, Physical Activity, and Stress Management Program | Wait-list Control | Total
Number analyzed (Participants) | 26 | 23 | 49
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.6 (4.20) | 47.7 (4.70) | 47.10 (4.50)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 23 | 49
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 26 | 23 | 49
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 26 | 23 | 49
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 26 | 23 | 49

OUTCOME MEASURES:

1. Primary Outcome: Change in Mean Systolic and Diastolic Blood Pressure (mm/Hg) From Baseline (Time 1) to Time 2
Description: Blood pressure will be measured in the right arm using a digital monitor. Participants will be seated comfortably with feet flat on the floor in a chair with back supported and the right arm resting on a table. The patient should be seated for 3-5 minutes without talking or moving around before recording the first blood pressure reading. Blood pressure will be repeated twice with the average computed. If it is not possible to measure blood pressure in the right arm, the left arm will be used and noted in the participant record.
Time Frame: Baseline (Time 1), Time 2 (Intervention completion, approximately 6 months)
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Education, Physical Activity, and Stress Management Program | Wait-list Control
Number analyzed (Participants) | 26 | 23
mmHg
  Systolic | -0.3 (2.7) | -2.4 (4.1)
  Diastolic | 1.2 (2.0) | 2.2 (2.7)

2. Primary Outcome: Change in Mean Systolic and Diastolic Blood Pressure From Baseline (Time 1) to Time 3
Description: as for outcome 1
Time Frame: Baseline (Time 1), Time 3 (6 month after completion of intervention, approximately 12 months)
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Education, Physical Activity, and Stress Management Program | Wait-list Control
Number analyzed (Participants) | 21 | 16
mmHg
  Systolic | 2.4 (3.3) | -2.8 (1.4)
  Diastolic | -1.0 (0.8) | -1.4 (1.4)

3. Primary Outcome: Change in Mean Arterial Stiffness From Baseline (Time 1) to Time 3
Description: Arterial stiffness will be measured by carotid-femoral pulse wave velocity and pulse wave analysis using the Vicorder® System (Skidmore Medical, Bristol, UK). Pulse wave velocity will be repeated twice with the average computed.
Time Frame: Baseline (Time 1), Time 3 (6 month after completion of intervention, approximately 12 months)
Measure: Mean (Standard Deviation); unit: meters per second (m/s)
Arm/Group | Education, Physical Activity, and Stress Management Program | Wait-list Control
Number analyzed (Participants) | 21 | 16
meters per second (m/s) | 0.0 (0.1) | -0.3 (1.1)

4. Primary Outcome: Changes in Mean Fasting Lipids (Total Cholesterol) From Baseline (Time 1) to Time 3
Description: Venous blood draw: A certified Research Assistant or Registered Nurse will perform a fasting blood draw. The participant will sit in a stationary chair with their arm of choice placed for the blood draw flat on the table, on top of the BloodBloc™ pad. The fasting blood sample will be analyzed by using the Cholestech LDX™ System at the Biobehavioral Laboratory in the School of Nursing at the University of North Carolina at Chapel Hill.
Time Frame: Baseline (Time 1), Time 3 (6 month after completion of intervention, approximately 12 months)
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Education, Physical Activity, and Stress Management Program | Wait-list Control
Number analyzed (Participants) | 21 | 16
mg/dL | 7.6 (11.7) | -13.9 (2.2)

5. Primary Outcome: Changes in Mean Fasting Lipids (Triglycerides) From Baseline (Time 1) to Time 3
Description: Venous blood draw: A certified Research Assistant or Registered Nurse will perform a fasting blood draw. The participant will sit in a stationary chair with their arm of choice placed for the blood draw flat on the table, on top of the BloodBloc pad. The fasting blood sample will be analyzed by using the Cholestech LDX™ System at the Biobehavioral Laboratory in the School of Nursing at the University of North Carolina at Chapel Hill.
Time Frame: Baseline (Time 1), Time 3 (6 month after completion of intervention, approximately 12 months)
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Education, Physical Activity, and Stress Management Program | Wait-list Control
Number analyzed (Participants) | 21 | 16
mg/dL | 15.4 (23.3) | -30.4 (16.0)

6. Primary Outcome: Changes in Mean Fasting Lipids (HDL Cholesterol) From Baseline (Time 1) to Time 3
Description: as for outcome 5
Time Frame: Baseline (Time 1), Time 3 (6 month after completion of intervention, approximately 12 months)]
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Education, Physical Activity, and Stress Management Program | Wait-list Control
Number analyzed (Participants) | 21 | 16
mg/dL | 3.89 (3.70) | -4.10 (2.20)

7. Primary Outcome: Changes in Mean Fasting Lipids (LDL Cholesterol) From Baseline (Time 1) to Time 3
Description: LDL Cholesterol will be computed at Time 1 and Time 3. Venous blood draw: A certified Research Assistant or Registered Nurse will perform a fasting blood draw. The participant will sit in a stationary chair with their arm of choice placed for the blood draw flat on the table, on top of the BloodBloc pad. The fasting blood sample will be analyzed by using the Cholestech LDX™ System at the Biobehavioral Laboratory in the School of Nursing at the University of North Carolina at Chapel Hill.
Time Frame: Baseline (Time 1), Time 3 (6 month after completion of intervention, approximately 12 months)
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Education, Physical Activity, and Stress Management Program | Wait-list Control
Number analyzed (Participants) | 21 | 16
mg/dL | 2.9 (9.8) | 5.4 (13.9)

8. Primary Outcome: Changes in Mean Fasting Glucose From Baseline (Time 1) to Time 3
Description: as for outcome 5
Time Frame: Baseline (Time 1), Time 3 (6 month after completion of intervention, approximately 12 months)
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Education, Physical Activity, and Stress Management Program | Wait-list Control
Number analyzed (Participants) | 21 | 16
mg/dL | 5.0 (2.3) | 9.9 (37.9)

9. Secondary Outcome: Change in Mean Weight (Kg) From Baseline (Time 1) to Time 2
Description: Weight will be measured twice using a digital scale placed on a hard, flat surface. The measurement will be recorded to the nearest 0.1-kg.
Time Frame: Baseline (Time 1), Time 2 (Intervention completion, approximately 6 months)
Measure: Mean (Standard Deviation); unit: Kg
Arm/Group | Education, Physical Activity, and Stress Management Program | Wait-list Control
Number analyzed (Participants) | 26 | 23
Kg | -2.9 (1.9) | -1.6 (0.7)

10. Secondary Outcome: Change in Mean Weight (Kg) From Baseline (Time 1) to Time 3
Description: as for outcome 9
Time Frame: Baseline (Time 1), Time 3 (6 month after completion of intervention, approximately 12 months)
Measure: Mean (Standard Deviation); unit: Kg
Arm/Group | Education, Physical Activity, and Stress Management Program | Wait-list Control
Number analyzed (Participants) | 21 | 16
Kg | -2.7 (1.4) | -2.1 (0.3)

11. Secondary Outcome: Change in Mean Body Mass Index (BMI) From Baseline (Time 1) to Time 2
Description: Participant weight and height will be used to calculate BMI. Calculation of BMI in kilograms divided by meters squared.
Time Frame: Baseline (Time 1), Time 2 (Intervention completion, approximately 6 months)
Measure: Mean (Standard Deviation); unit: Kg/m^2
Arm/Group | Education, Physical Activity, and Stress Management Program | Wait-list Control
Number analyzed (Participants) | 26 | 23
Kg/m^2 | -1.3 (5.4) | -0.2 (5.5)

12. Secondary Outcome: Change in Mean Body Mass Index (BMI) From Baseline (Time 1) to Time 3
Description: Participant weight and height will be used to calculate BMI. Calculation of BMI in kilograms divided by meters squared.
Time Frame: Baseline (Time 1), Time 3 (6 month after completion of intervention, approximately 12 months)
Measure: Mean (Standard Deviation); unit: Kg/m^2
Arm/Group | Education, Physical Activity, and Stress Management Program | Wait-list Control
Number analyzed (Participants) | 21 | 16
Kg/m^2 | -1.3 (0.3) | -0.9 (5.9)

13. Secondary Outcome: Change in Mean Adiposity (Waist Circumference) From Baseline (Time 1) to Time 2
Description: Waist circumference will be measured at the level of the umbilicus in centimeters using a measuring tape.
Time Frame: Baseline (Time 1), Time 2 (Intervention completion, approximately 6 months)
Measure: Mean (Standard Deviation); unit: centimeters (cm)
Arm/Group | Education, Physical Activity, and Stress Management Program | Wait-list Control
Number analyzed (Participants) | 26 | 23
centimeters (cm) | -6.0 (4.6) | -5.4 (1.4)

14. Secondary Outcome: Change in Mean Adiposity (Waist Circumference) From Baseline (Time 1) to Time 3
Description: Waist circumference will be measured at the level of the umbilicus in centimeters using a measuring tape.
Time Frame: Baseline (Time 1), Time 3 (6 month after completion of intervention, approximately 12 months)
Measure: Mean (Standard Deviation); unit: centimeters (cm)
Arm/Group | Education, Physical Activity, and Stress Management Program | Wait-list Control
Number analyzed (Participants) | 21 | 16
centimeters (cm) | -2.9 (0.4) | -1.6 (1.2)

15. Secondary Outcome: Change in Proportion of Participants Meeting Recommended Intake of Fruits, Vegetables and Fish (Food Behavior Checklist) Baseline (Time 1) to Time 2
Description: Change in proportion of participants meeting American Heart Association-recommended intake of each of the following: fruits, vegetables, and fish based on completing the Food Behavior Checklist. The Food Behavior Checklist asks participants to indicate the number of daily servings consumed for each category..
Time Frame: Baseline (Time 1), Time 2 (Intervention completion, approximately 6 months)
Measure: Number; unit: proportion of participants
Arm/Group | Education, Physical Activity, and Stress Management Program | Wait-list Control
Number analyzed (Participants) | 26 | 23
proportion of participants
  Fruit | 0.0 | 0.044
  Vegetable | 0.038 | 0.043
  Fish | 0.077 | -0.044

16. Secondary Outcome: Change in Proportion of Participants Meeting Recommended Intake of Fruits, Vegetables and Fish (Food Behavior Checklist) Baseline (Time 1) to Time 3
Description: as for outcome 15
Time Frame: Baseline (Time 1), Time 3 (6 month after completion of intervention, approximately 12 months)
Measure: Number; unit: proportion of participants
Arm/Group | Education, Physical Activity, and Stress Management Program | Wait-list Control
Number analyzed (Participants) | 21 | 16
proportion of participants
  Fruit | 0.076 | 0.043
  Vegetable | 0.153 | 0.043
  Fish | 0.115 | -0.174

17. Secondary Outcome: Change in Health Behaviors (Accelerometer Measurement for 7 Days) From Baseline (Time 1) to Time 2
Description: The participant will wear an accelerometer for 7 days total. This information will be uploaded into the computer to provide data on low, moderate, and high intensity physical activity. The proportion of participants across categories will be reported.
Time Frame: Baseline (Time 1), Time 2 (Intervention completion, approximately 6 months)
Population: No data were collected for this outcome. Due to the COVID-19 pandemic many of the community-based organizations that were going to serve as pick-up and drop-off for the accelerometers were closed. In addition, the funding source for purchasing accelerometers was lost.
Arm/Group | Education, Physical Activity, and Stress Management Program | Wait-list Control
Number analyzed (Participants) | 0 | 0

18. Secondary Outcome: Change in Health Behaviors (Accelerometer Measurement for 7 Days) From Baseline (Time 1) to Time 3
Description: as for outcome 17
Time Frame: Baseline (Time 1), Time 3 (after 6 months with no contact from the study staff, approximately 12 months)
Population: as for outcome 17
Arm/Group | Education, Physical Activity, and Stress Management Program | Wait-list Control
Number analyzed (Participants) | 0 | 0

19. Secondary Outcome: Change in Median Eating Self-Efficacy Questionnaire From Baseline (Time 1) to Time 2
Description: This is a 25-item questionnaire asking how much difficulty the participant has with controlling her eating in social situations and every day. The range of scores go from 1 to 7 with 1 being no difficulty controlling eating to 4 moderate difficulty controlling eating to 7 the most difficulty controlling eating. The 25 questions are added to produce a total score (0-175). A lower score equals less difficulty controlling eating and a higher score equals more difficulty controlling eating.
Time Frame: Baseline (Time 1), Time 2 (Intervention completion, approximately 6 months)
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Education, Physical Activity, and Stress Management Program | Wait-list Control
Number analyzed (Participants) | 26 | 23
score on a scale | -7.5 [-37 to 86.25] | -35.0 [-62 to 84.5]

20. Secondary Outcome: Change in Median Eating Self-Efficacy Questionnaire From Baseline (Time 1) to Time 3
Description: as for outcome 19
Time Frame: Baseline (Time 1), Time 3 (after 6 months with no contact from the study staff, approximately 12 months)
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Education, Physical Activity, and Stress Management Program | Wait-list Control
Number analyzed (Participants) | 21 | 16
score on a scale | -11.0 [-37 to 49.25] | 31.0 [1.0 to 54.0]

21. Secondary Outcome: Change in Mean Exercise Self-Efficacy Questionnaire From Baseline (Time 1) to Time 2
Description: This is a 9-item questionnaire asking how much confidence the participant has doing particular exercises. The range of scores go from 0 to 10 with 0 being she is not confident at all (low self-efficacy) and and 10 being that she is certain she can do it (high self-efficacy). The numbers are summed for a total score (0-90) with higher scores indicating greater exercise self-efficacy.
Time Frame: Baseline (Time 1), Time 2 (Intervention completion, approximately 6 months)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Education, Physical Activity, and Stress Management Program | Wait-list Control
Number analyzed (Participants) | 26 | 23
score on a scale | -0.5 (2.1) | -2.4 (2.3)

22. Secondary Outcome: Change in Mean Exercise Self-Efficacy Questionnaire From Baseline (Time 1) to Time 3
Description: as for outcome 21
Time Frame: Baseline (Time 1), Time 3 (after 6 months with no contact from the study staff, approximately 12 months)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Education, Physical Activity, and Stress Management Program | Wait-list Control
Number analyzed (Participants) | 21 | 16
score on a scale | -10.4 (3.3) | -4.9 (3.0)

23. Secondary Outcome: Change in Mean Sleep Quality Questionnaire From Baseline (Time 1) to Time 2
Description: This is a 4-item question questionnaire previously used in studies during the menopause transition. Each question is scored from 0 to 4, with 0 being indicating no difficulty with sleep in the past two weeks and 4 indicating five or more times a week of difficulty sleeping. The numbers are summed for a total score (0-16). A lower number indicates that the participant does not have difficulty sleeping and a higher number means that the participant has a lot of difficulty sleeping.
Time Frame: Baseline (Time 1), Time 2 (Intervention completion, approximately 6 months) ]
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Education, Physical Activity, and Stress Management Program | Wait-list Control
Number analyzed (Participants) | 26 | 23
score on a scale | -2.1 (4.1) | 0.4 (4.9)

24. Secondary Outcome: Change in Mean Sleep Quality Questionnaire From Baseline (Time 1) to Time 3
Description: as for outcome 23
Time Frame: Baseline (Time 1), Time 3 (after 6 months with no contact from the study staff, approximately 12 months)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Education, Physical Activity, and Stress Management Program | Wait-list Control
Number analyzed (Participants) | 21 | 16
score on a scale | -2.5 (4.1) | -1.5 (4.9)

25. Secondary Outcome: Change in Median High-Sensitivity C-Reactive Protein From Baseline (Time 1) to Time 3
Description: Serum high-sensitivity C-reactive protein levels will by obtained by from a fasting blood sample and at the Biobehavioral Laboratory in the School of Nursing at the University of North Carolina at Chapel Hill.
Time Frame: Baseline (Time 1), Time 3 (after 6 months with no contact from the study staff, approximately 12 months)
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | Education, Physical Activity, and Stress Management Program | Wait-list Control
Number analyzed (Participants) | 21 | 16
ng/mL | 86.6 [45.2 to 404.6] | 272.3 [31.6 to 372.2]

26. Secondary Outcome: Change in Mean Hair Cortisol Levels From Baseline (Time 1) to Time 3
Description: Cortisol will be obtained from hair samples and analyzed using a standard laboratory protocol at the Biobehavioral Laboratory in the School of Nursing at the University of North Carolina at Chapel Hill.
Time Frame: Baseline (Time 1), Time 3 (after 6 months with no contact from the study staff, approximately 12 months)
Measure: Mean (Standard Deviation); unit: pg/mg
Arm/Group | Education, Physical Activity, and Stress Management Program | Wait-list Control
Number analyzed (Participants) | 21 | 16
pg/mg | 24.29 (89.05) | 13.39 (29.01)

27. Secondary Outcome: Number of Eligible Women That Agree to Participate in the Study
Description: This will be defined as a number of women that agree to participate in the study out of the total women screened for the study.
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Groups:
- Total Participants Screened: This is the total number of participants that were screened for eligibility.
Arm/Group | Total Participants Screened
Number analyzed (Participants) | 143
Participants | 49

28. Secondary Outcome: Time for Recruitment
Description: This will be defined as time (days) from initial contact with research staff to randomization into the study.
Time Frame: Baseline
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Education, Physical Activity, and Stress Management Program | Wait-list Control
Number analyzed (Participants) | 26 | 23
days | 30 [30 to 105] | 90 [45 to 121.5]

29. Secondary Outcome: Mean Proportion of Group Sessions Participants Attend
Description: The attendance rate will be defined as the proportion of group sessions the participant attends.The mean proportion of sessions that participants attended out of the total of 15 sessions offered is reported.
Time Frame: Time 2 (Intervention completion, approx. 6 months)
Population: This only applies to the intervention arm because the Wait-list Control arm did not have any sessions to attend during the study.
Measure: Mean (Standard Deviation); unit: proportion of sessions attended
Arm/Group | Education, Physical Activity, and Stress Management Program | Wait-list Control
Number analyzed (Participants) | 26 | 0
proportion of sessions attended | 0.533 (1.0) |

30. Secondary Outcome: Number of Participants at Post-intervention (Time 2) and Study Completion (Time 3)
Description: The retention rate will be defined as the percentage of participants remaining in the study at post-intervention and at study completion.
Time Frame: Time 2 (Intervention completion, approx. 6 months) and Time 3 (after 6 months with no contact from the study staff, approximately 12 months)
Measure: Count of Participants; unit: Participants
Arm/Group | Education, Physical Activity, and Stress Management Program | Wait-list Control
Number analyzed (Participants) | 26 | 23
Participants
  Post-intervention (Time 2) | 22 | 20
  Study Completion (Time 3) | 21 | 16

31. Secondary Outcome: Proportion of Participants That Attend at Least 80% of the Intervention Session (12-15 Sessions).
Description: A Research Assistant will assess fidelity of the intervention fidelity by keeping an attendance log.
Time Frame: Time 2 (Intervention completion, approx. 6 months)
Population: This is outcome is only applicable to the intervention group.
Measure: Number; unit: proportion of participants
Arm/Group | Education, Physical Activity, and Stress Management Program | Wait-list Control
Number analyzed (Participants) | 26 | 0
proportion of participants | 0.26923077 |

32. Secondary Outcome: Number of Participants That Would Recommend the Study to a Friend or Relative.
Description: Participants will be asked: "If a friend or relative were to be asked to take part in the study, how likely would you be to recommend that they participate?"
Time Frame: Time 3 (after 6 months with no contact from the study staff, approximately 12 months)
Measure: Count of Participants; unit: Participants
Arm/Group | Education, Physical Activity, and Stress Management Program | Wait-list Control
Number analyzed (Participants) | 21 | 16
Participants | 20 | 15

33. Other Pre Specified Outcome: Change in Proportion of Participants Reporting Vasomotor Symptoms From Baseline (Time 1) to Time 2
Description: Participants will report experiencing any vasomotor symptoms (night sweats, hot flashes) in the past two weeks
Time Frame: Baseline (Time 1), Time 2 (Intervention completion, approximately 6 months)
Measure: Number; unit: proportion of participants
Arm/Group | Education, Physical Activity, and Stress Management Program | Wait-list Control
Number analyzed (Participants) | 26 | 23
proportion of participants | -0.193 | -0.305

34. Other Pre Specified Outcome: Change in Proportion of Participants Reporting Vasomotor Symptoms From Baseline (Time 1) to Time 3
Description: Participants will report experiencing any vasomotor symptoms (night sweats, hot flashes) in the past two weeks.
Time Frame: Baseline (Time 1), Time 3 (after 6 months with no contact from the study staff, approximately 12 months)
Measure: Number; unit: proportion of participants
Arm/Group | Education, Physical Activity, and Stress Management Program | Wait-list Control
Number analyzed (Participants) | 21 | 16
proportion of participants | -0.154 | -0.261

ADVERSE EVENTS:
Time Frame: From the time of signing informed consent through study completion, a total of approximately 18 months.
Description: Adverse events were collected throughout the duration of the study (i.e., Baseline through Month 12). Although Wait-list control participants were offered the opportunity to receive education sessions after all participants had completed Month 12 visits and the study was closed, this occurred after study completion and outside of the scope of the study. Thus, no adverse events were collected for Wait-list control participants who decided to receive education sessions after study completion.
Arm/Group | Education, Physical Activity, and Stress Management Program | Wait-list Control
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/23
Other Adverse Events (participants affected / at risk) | 0/26 | 0/23

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-08-09): https://cdn.clinicaltrials.gov/large-docs/51/NCT04313751/Prot_SAP_001.pdf
  • Informed Consent Form (2020-12-23): https://cdn.clinicaltrials.gov/large-docs/51/NCT04313751/ICF_000.pdf